CLINICAL TRIAL: NCT02807194
Title: Epidural Anesthesia Versus General Anesthesia for Elective Lumbar Disk Surgery in a Outpatient Basis
Brief Title: Ambulatory Lumbar Disk Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PO13123
Record Dates: First submitted 2016-06-16; First posted 2016-06-21 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Lumbar Disk Surgery
MeSH Terms: interventions — Anesthesia, Spinal; Anesthesia, General

ARMS (2):
- general anesthesia (Experimental): 'lumbar disc herniation'
  Interventions: Other: general anesthesia; Procedure: lumbar disc herniation
- spinal anesthesia (Experimental): 'lumbar disc herniation'
  Interventions: Other: spinal anesthesia; Procedure: lumbar disc herniation

INTERVENTIONS:
Other: spinal anesthesia
  Arms: spinal anesthesia
Other: general anesthesia
  Arms: general anesthesia
Procedure: lumbar disc herniation

SUMMARY:
Primary Goal: To compare the clinical outcomes of spinal anesthesia and general anesthesia in surgery for lumbar disc herniation.

DETAILED DESCRIPTION:
Patients included: All patients in the neurosurgery department of the University Hospital of Reims or in the neurosurgery department of CHG Chalons en Champagne for surgical management of lumbar disc herniation and agreeing to participate in the research. The types of anesthesia (general anesthesia or spinal anesthesia) will be randomized.

Investigation Plan: Participation in the research will be available to any eligible patient during the anesthesia consultation prior hospitalization for surgery. If the patient agrees to participate in research, randomization of the anesthetic technique will be realized. The anesthetist and the patient will be informed of the outcome of this randomization. Hospitalization of patients will not be changed. They will be hospitalized in inpatient, as usual, with an entry the day before surgery and an outlet the next day (without complications). The surgery itself will not be changed. The patient's postoperative monitoring will not be changed. Data will be collected for each patient: demographic data, medical data, data about the intervention and anesthesia, postoperative data management.

ELIGIBILITY:
Inclusion Criteria:

* single lumbar disk herniation elective for surgery

Exclusion Criteria:

* Patients with haemostatic disorder
* Patients with lumbar spine surgery history
* Patients with sciatica called "hyperalgesia" resistant to treatment including systemic corticosteroids and 3 WHO bearing analgesics (oral morphine)
* Patients with true paralyzing sciatica with motor disorders compatible with the path of the root compressed by the herniation
* Patients with sphincter disorders
* Patients with herniated disc multistage
* Pregnant women
* Patients with comorbid against-showing the elongated position, including cardiorespiratory comorbidities
* Minors patients
* Patients protected by law.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-03; Primary Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
consumption of analgesic Level III (according to WHO criteria) | 24hours

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, France, Reims, France